CLINICAL TRIAL: NCT03792178
Title: Evaluation of Post-operative Sensitivity of Bulk Fill Resin Composite Versus the Nano Resin Composite.
Acronym: EPSBN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rasmia Mamdouh Ali Salem (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Rasmia Mamdouh Ali Salem, Assistant lecturer at operative Department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 150405
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Sensitivity
Keywords: Post operative sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: bulk fill resin composite placement techqniues versus nano resin composite at postoperative hypersensitivity
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nano resin composite (Active Comparator): are types of synthetic resins which are used in dentistry as restorative material or adhesives.
  Interventions: Other: Bulk fill composite; Other: Nano resin composite
- Bulk fill composite (Experimental): Bulk- ll composites are claimed to be restorative materials used in deep preparations and effectively photoactivated in layers up to 4 mm.
  Interventions: Other: Bulk fill composite; Other: Nano resin composite

INTERVENTIONS:
Other: Bulk fill composite — Composite resin dental material
Other: Nano resin composite — Dental composite material

SUMMARY:
Our study evaluated and compared the postoperative sensitivity of the placement technique (incremental and bulk fill) in class II posterior composite resin restorations bonded with two different adhesive strategies (self-etch and etch-and-rinse).Sixty patients were randomly selected, their age range from 25 to 40 years old. They were divided into 2 main groups according to the packing technique of composite material; incremental Tetric Evoceram and Tetric Evoceram bulk fill composite.30 patients (n=30) were selected for incremental Tetric Evoceram composite restorations and they were equally divided according to the adhesive systems used (etch and rinse or self-etch adhesive strategy) (n=15 teeth).30 patients (n=30) were selected for Tetric Evoceram bulk fill composite restorations and they were equally divided according to the adhesive systems used (etch and rinse or self-etch adhesive strategy) (n=15 teeth).Post-operative pain assessed at 24 hours, 1 week and 1 month using the visual Analog Scale Score (VAS).Each patient was instructed to place a vertical mark on the VAS line at home to indicate the intensity of pain at each assessment period.

DETAILED DESCRIPTION:
Our results revealed that when the two composite types using self-etch adhesive system & total-etch adhesive system were evaluated; there was no statistically significant difference between the two composite types after 1 day, 1 week as well as 1 month.

When the two adhesive systems were compared using Bulk Fill composite & incremental Nano resin composite there was no statistically significant difference between the two adhesive systems after 1 day, 1 week as well as 1 month.

Using Bulk Fill composite with self-etch adhesive; there was a statistically significant decrease in prevalence of hypersensitivity after 1 week. There were no cases with hypersensitivity after 1 week as well as 1 month. Using Bulk Fill composite with Total etch adhesive; there was a statistically significant decrease in prevalence of hypersensitivity after 1 week as well as from 1 week to 1 month.

Using Incremental Nano resin composite with self-etch adhesive; there was a statistically significant decrease in prevalence of hypersensitivity after 1 week as well as from 1 week to 1 month. Using Incremental Nano resin composite with Total etch adhesive; there was a statistically significant decrease in prevalence of hypersensitivity after 1 week as well as from 1 week to 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients must show no signs of spontaneous dental or orofacial pain.
* The presence of molar and premolar class II teeth requiring composite restorations for the treatment of primary carious lesions
* The selected teeth should have an occlusal contact with natural or crowned antagonist teeth
* The selected teeth should have a proximal contact with the adjacent teeth.
* Shallow and mid-sized cavity depths will be included in the study .

Exclusion Criteria:

* Increasing pre-operative sensitivity of the selected teeth.
* Teeth with abnormal periapical anatomy or caries that will be likely to result in very deep restorations.
* Teeth with old restorations or severely destructed dental crowns.
* Teeth with spontaneous pain
* Tempro-mandibular joint problems involving symptomatic pain.
* Patients taking analgesics that could alter their normal pain perception level.
* Pregnancy or breast feeding, acute and chronic systemic diseases, immunecompromised patients.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
sensitivity | one month follow up
  post operative sensitivity

IPD SHARING:
Plan to Share IPD: Undecided